CLINICAL TRIAL: NCT05244473
Title: A Phase 1, Single-blind, Dose-escalation Study to Assess the Safety and Tolerability of Brentuximab Vedotin (ADCETRIS®) in Subjects With Human Immunodeficiency Virus (HIV)
Brief Title: A Safety Study of Brentuximab Vedotin in Participants With HIV
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn due to low patient accrual.
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGN35-035
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Immunological Nonresponder; Seattle Genetics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Brentuximab Vedotin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brentuximab vedotin + ART (Experimental): Brentuximab vedotin given on Day 1 and Day 15. ART will be given throughout the study.
  Interventions: Drug: brentuximab vedotin; Drug: ART
- Placebo + ART (Placebo Comparator): Placebo given on Day 1 and Day 15. ART will be given throughout the study.
  Interventions: Drug: Placebo; Drug: ART

INTERVENTIONS:
Drug: brentuximab vedotin — Given into the vein (IV; intravenously)
  Other Names: ADCETRIS
  Arms: Brentuximab vedotin + ART
Drug: Placebo — Given by IV
  Arms: Placebo + ART
Drug: ART — Daily use of a combination of HIV medicines

SUMMARY:
This study will test brentuximab vedotin to see if it is safe for people with human immunodeficiency virus (HIV) who have low CD4+ and have received antiretroviral therapy (ART) treatment. It will also see if brentuximab vedotin raises CD4+ counts. It will study the side effects of this drug as well. A side effect is anything a drug does to the body besides treating the disease.

In this study participants will be assigned randomly to a group. Participants will get either brentuximab vedotin or placebo. A placebo looks like the drug but does not contain any medicine in it. All participants will keep getting ART during the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive with documentation of infection
* Immunological nonresponder, defined as:

  * Has been on ART with an HIV viral load <50 copies/mL for at least 24 months
  * Has a CD4+ T-cell lymphocyte count between 51 to 200 cells/µL
* Life expectancy of >9 months.
* Participant is negative for hepatitis B, or if infected with hepatitis B, receiving anti-hepatitis B therapy
* Participants with a history of hepatitis C virus (HCV) are eligible if they have completed therapy for HCV and show sustained virologic remission (12 weeks or more)

Exclusion Criteria:

* Any currently active AIDS-defining illness per Category C conditions according to the CDC Classification System for HIV Infection, with the following exceptions:

  * Limited cutaneous Kaposi's sarcoma not currently requiring systemic therapy
  * Wasting syndrome due to HIV or any other AIDS-defining illness for which no therapeutic treatment is required OR the required treatment is not included in the list of prohibited medications
* Acute liver disease or any other active infection secondary to HIV requiring acute therapy
* History of progressive multifocal leukoencephalopathy (PML)
* Prior clinical John Cunningham virus (JCV) infection, history of JCV identified in cerebrospinal fluid, or presence of JCV antibodies at screening
* Cirrhosis secondary to any cause
* Any immunomodulating therapy (excluding premedication steroid) within 4 weeks prior to the screening visit
* Prior malignancy within 2 years other than cutaneous basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, anal intraepithelial neoplasia, or cutaneous Kaposi's sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30 days after last study treatment
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment
Number of participants with laboratory abnormalities | Approximately 1 year
Number of participants with dose-limiting toxicities (DLTs) by dose level | Up to 30 days

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) | Approximately 4 months
  Pharmacokinetic (PK) Parameter
Maximum concentration (Cmax) | Approximately 4 months
  PK Parameter
Time to maximum concentration (Tmax) | Approximately 4 months
  PK Parameter
Apparent terminal half-life (t1/2) | Approximately 4 months
  PK Parameter
Trough concentration (Ctrough) | Approximately 4 months
  PK Parameter
Incidence of antidrug antibodies (ADAs) | Approximately 4 months
Proportion of participants with CD4+ T-cell lymphocyte count >200 cells/µL | Approximately 1 year
Proportion of participants with CD4+ T-cell lymphocyte count >200 cells/µL, with a minimum increase of 50 cells/µL | Approximately 1 year
Duration of CD4+ T-cell lymphocyte count increases >200 cells/µL | Approximately 1 year
  The time from start of the first occurrence of CD4+ T-cell count increases to the level >200 cells/µL to the first occurrence of CD4+ T-cell count to the level <200 cells/µL
Duration of CD4+ T-cell lymphocyte count increases >200 cells/µL with a minimum increase of 50 cells/µL | Approximately 1 year
  The time from start of the first occurrence of CD4+ T-cell count increases to the level >200 cells/µL to the first occurrence of CD4+ T-cell count to the level <200 cells/µL with a minimum increase of 50 cells/µL
Change from baseline in CD4+ T-cell lymphocyte counts | Approximately 1 year
  The change from baseline in CD4+ T-cell lymphocyte counts will be summarized based on observed values.
Change from baseline in CD4+ T cell percentage | Approximately 1 year
  The change from baseline in CD4+ T cell percentage will be summarized based on observed values.
Change from baseline in CD8+ T-cell lymphocyte counts | Approximately 1 year
  The change from baseline CD8+ T-cell lymphocyte counts will be summarized based on observed values.
Change from baseline in CD4:CD8 ratio | Approximately 1 year
  The change from baseline in CD4:CD8 ratio will be summarized.
Change from baseline in Treg and other T-cell subsets | Approximately 6 months
Proportion of subjects with HIV viral load <50 copies/mL | Approximately 1 year
  The proportion of subjects with HIV viral load <50 copies/mL will be summarized.
Proportion of subjects with fatal or non-fatal acquired immunodeficiency syndrome (AIDS) related opportunistic disease or death from any cause | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Shustov, MD, Study Director — Seagen Inc.
Locations (2):
- United States (2):
  - University of California at San Francisco, San Francisco, California
  - University of Illinois at Chicago, Chicago, Illinois